CLINICAL TRIAL: NCT07277738
Title: Precision Supplemental Imaging in Women With Dense Breasts (PSID Trial)
Brief Title: Precision Supplemental Imaging in Women With Dense Breasts
Acronym: PSID
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 202511123
Record Dates: First submitted 2025-12-02; First posted 2025-12-11 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer; Cancer of the Breast
Keywords: Dense breasts; Abbreviated MRI; Risk assessment
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammography; Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: The feasibility study will enroll 78 evaluable women and will be sequential enrollment. The sample size for the randomized controlled portion of this study will depend on the results of the feasibility portion of the study and it will be parallel enrollment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Feasibility: Recommended MRI (Experimental): Consenting and eligible participants will be recommended to undergo MRI and will be followed to determine whether they complete the MRI.
  Interventions: Device: Prognosia Breast; Device: Mammogram; Device: MRI
- Arm A: Intervention - MRI + subsequent annual screening mammogram with MRI (Experimental): Consenting and eligible participants will undergo an MRI and subsequent annual screening mammogram with MRI.
  Interventions: Device: Prognosia Breast; Device: Mammogram; Device: MRI
- Arm B: Regular Care - annual screening mammogram (Active Comparator): Consenting and eligible participants will undergo annual screening mammogram per standard of care.
  Interventions: Device: Mammogram

INTERVENTIONS:
Device: Prognosia Breast — The risk output from this algorithm is calibrated to US Surveillance, Epidemiology, and End Results (SEER) 5-year risk and so estimates for each woman the personal 5-year risk.
  Other Names: MRS; Mammogram absolute risk score
  Arms: Arm A: Intervention - MRI + subsequent annual screening mammogram with MRI; Feasibility: Recommended MRI
Device: Mammogram — Standard of care annual screening mammogram
Device: MRI — MRI at the time of annual screening mammogram
  Other Names: Magnetic resonance imaging
  Arms: Arm A: Intervention - MRI + subsequent annual screening mammogram with MRI; Feasibility: Recommended MRI

SUMMARY:
Recent research has shown that, among women with extremely dense breasts and normal results on mammogram, magnetic resonance imaging (MRI) use has significantly reduced the occurrence of breast cancer that is diagnosed during the time between two regular screening mammograms (also known as interval cancers).

The investigators have developed and validated an approach to use the whole mammogram image, develop a mammogram risk score (MRS), and calibrate this to the SEER breast cancer incidence rates for US women. This model (Prognosia Breast) generates an absolute 5-year risk of breast cancer and classifies approximately 5.7% of the population as high risk using the ASCO 3% cut point as used for endocrine therapy to reduce risk. Follow-up generates an incidence of 25.2 cases per 1,000 women per year.

ELIGIBILITY:
Inclusion Criteria:

* Normal screening mammogram within 90 days prior to enrollment.
* Dense breasts, either:

  * Class C density ("the breasts are heterogeneously dense, which may obscure small masses")
  * Class D density ("the breasts are extremely dense, which lowers the sensitivity of mammography")
* MRS risk estimate at > 3% 5-year risk of breast cancer.
* Female.
* Between 25 and 55 years of age (inclusive).
* Ability to understand and willingness to sign an IRB approved written informed consent document.

Exclusion Criteria:

* More than 1 prior mammogram
* Contraindication to MRI with contrast (e.g. claustrophobia, metal objects in the body, known sensitivity/allergy to gadolinium).
* Prior or concurrent malignancy whose natural history has the potential to interfere with the study intervention (breast cancer or LCIS). Patients with prior or concurrent malignancy that does NOT meet that definition are eligible for this trial.
* Prior MRI screening of the breast.
* Known to be BRCA 1/2 positive or presence of any other known high penetrance genetic marker.
* Is receiving any chemoprevention.
* Has breast implants.
* Is breastfeeding.

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of successful recommendations for MRI (Feasibility portion only) | Through completion of follow-up (estimated to be 24 months)
  Successful recommendation of MRI is defined as completion of MRI by women referred for MRI.
2-year detection rate (Randomized Controlled Trial only) | 2 years
  Events including interval breast cancer or invasive breast cancer of a size ≥15mm or being lymph node positive, by arm

SECONDARY OUTCOMES:
Sample size for randomized controlled trial (Feasibility portion only) | Through completion of follow-up (estimated to be 24 months)
  At the completion of the feasibility study, the investigators will use the feasibility study data to inform and calculate the sample size for the subsequent randomized 2-arm trial, and if feasible and results are promising, the investigators will propose a randomized 2-arm trial to evaluate the effectiveness of MRI screening in terms of 2-year event rate.
Number and percentage of recalls (Feasibility portion only) | Through completion of follow-up (estimated to be 24 months)
Positive predictive value for recall for additional testing and biopsy (Feasibility portion only) | Through completion of follow-up (estimated to be 24 months)
Number and percentage of recalls (Randomized Controlled Trial only) | Through completion of follow-up (estimated to be 24 months)
Positive predictive value for recall for additional testing and biopsy (Randomized Controlled Portion only) | Through completion of follow-up (estimated to be 24 months)

CONTACTS AND LOCATIONS:
Overall Officials: Tabassum Ahmad, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Proposals should be directed to the Principal Investigator. To gain access, data requestors will need to sign a data access agreement and provide a methodologically sound proposal.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu